CLINICAL TRIAL: NCT03699852
Title: Characterization of the Repair Process and the Effects of Photobiomodulation in a Donor Area of Partial Thickness Skin Graft After Burn
Brief Title: Effect of Photobiomodulation in a Partial Thickness Autogenous Skin Graft Donor Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rosadélia
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Healing Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED group (Experimental): The study had two groups of participants: the LED group (GL) and the control group (GC), both with Membracel®, a porous membrane that regenerates crystalline cellulose, as the primary cover in the donor area of the skin graft (no secondary cover was used) ). In one of the groups (GL), a light-emitting diode (LED) plate was applied, which was covered with sterile waterproof and transparent film to prevent contamination. The participant was positioned so that the skin graft donor area was accessible. The LED plate covered the entire skin donor area and was irradiated with a radiant exposure of 1.53J / cm2 and irradiance of 2.55 mW / cm2 for 10 minutes. The LED plate was applied in contact with the skin graft donor area in the immediate postoperative period and on Membracel® on the 1st, 3rd, 5th and 7th postoperative days. The primary coverage remained until spontaneous removal.
  Interventions: Radiation: Membracel and LED photobiomodulation
- Control group (Other): The participants remained and were evaluated under the same conditions. The only difference between the groups is that no LED photobiomodulation session was applied to the control group.
  Interventions: Other: Membracel

INTERVENTIONS:
Radiation: Membracel and LED photobiomodulation — Participants were positioned so that the skin graft donor area was accessible. A light-emitting diode (LED) plate was covered with sterile transparent and waterproof film to prevent contamination when in contact with the donor area. The application was in contact, with full coverage of the surgical wound and was irradiated with radiant exposure of 1.53J / cm2 and irradiance of 2.55 mW / cm2 for 10 minutes. It is worth mentioning that the LED plate was applied in direct contact with the skin graft donor area in the immediate postoperative period and on the primary cover used (Membracel®) on the 1st, 3rd, 5th and 7th postoperative days. Coverage remained until spontaneous departure. The researcher and the participants used specific goggles for this procedure.
  Arms: LED group
Other: Membracel — This group did not receive LED application, remaining with the skin donor area covered by Membracel® and were evaluated under the same conditions.
  Arms: Control group

SUMMARY:
This is a clinical study with a controlled series of cases, whose objectives were: to evaluate the effects of FBM, using LED, on the repair process of the skin graft donor area treated with Membracel® and LED versus Membracel ®; to evaluate the evolution of the quality of the aspects of the skin donor area, through the score obtained by the modified Bates-Jensen Scale; the intensity of the pain reported by the participants; the size of the wound area until the 7th postoperative (PO) period and the time for re-epithelialization of the donor area. Data collection was performed at the Burn Unit of the General Hospital "Dr. José Pangella", from Vila Penteado, São Paulo, Brazil. The sample consisted of 21 participants and 25 donor areas, 13 of which were from the control group, which received only conventional treatment (Membracel®) and 12 from the experimental group: Membracel® and LED. Data collection instruments were used: medical records of the participants, anamnesis and physical examination, the scales: pain (Visual Analogic Scale - VAS) and Bates-Jensen to accompany the re-epithelialization process and the measurement of donor skin areas in the postoperative period. Quantitative variables were represented by the mean, standard deviation and the median and interquartile range. The comparison of the distributions of these variables between groups was performed using the Mann-Whitney test.

DETAILED DESCRIPTION:
The use of FBM, showing beneficial effects on wounds, is well described in the literature. The reported findings include anti-inflammatory action, better tissue organization, acceleration of angiogenesis, stimulation of leukocyte chemotaxis and reduction of donor area size in animals and humans. This is a clinical study with a controlled series of cases, whose objectives were: to evaluate the effects of FBM, using LED, on the repair process of the skin graft donor area treated with Membracel® and LED versus Membracel ®; to evaluate the evolution of the quality of the aspects of the skin donor area, through the score obtained by the modified Bates-Jensen Scale; the intensity of the pain reported by the participants; the size of the wound area until the 7th postoperative (PO) period and the time for re-epithelialization of the donor area. Data collection was performed at the Burn Unit of the General Hospital "Dr. José Pangella", from Vila Penteado, São Paulo, Brazil, from December 2018 to January 2020. The sample consisted of 21 participants and 25 donor areas, 13 of which were from the control group, which received only conventional treatment (Membracel®) and 12 from the experimental group: Membracel® and LED. Data collection instruments were used: medical records of the participants, anamnesis and physical examination, the scales: pain (Visual Analogic Scale - VAS) and Bates-Jensen to accompany the re-epithelialization process and the measurement of donor skin areas in the postoperative period. Participants were identified by Arabic numbers, according to the order of arrival at the Hospital. Quantitative variables were represented by the mean, standard deviation and the median and interquartile range. The comparison of the distributions of these variables between groups was performed using the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with burns requiring a partial thickness skin graft from a healthy donor area;
* Both sexes;
* Aged 18 years or older;
* Regardless of skin color or comorbidities.

Exclusion Criteria:

* Patients with a full-thickness skin donor area;
* Under the age of 18;
* Those who refuse to participate;
* With infected wounds that evolved with purulent exudation during treatment;
* Cancer participants treated with radiation therapy or chemotherapy;
* With systemic infection;
* Corticosteroid use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in the Bates-Jensen Wound Assessment Tool (BWAT) | Every two days until wound reepithelialization
  This scale evaluates size, depth, edges, detachment, type and amount of necrotic tissue, type and amount of exudate, edema and hardening of the peripheral tissue, skin color around the wound, granulation tissue and epithelization. The measurement scale is of the Likert type, with five points, with 1 indicating the best condition of the wound and 5, the worst condition. The total score is obtained with the sum of all the items and can vary from 13 to 65 points, with the highest scores indicating the worst conditions of the wound. The items: size, depth, edges, and detachment should be scored with zero when the lesions are healed. The instrument contains two items: location and form - which are not part of the total score.
Change in the Analogic visual scale | Every two days, until the 7th day after the procedure.
  The scale allows for "validation" by the participant, as he or she experiences pain and is therefore an expert on the pain pattern, location, intensity and nature.
Time for donor area reepithelialization | Once a week
  The LED Group and Control Group donor areas were evaluated for time to reepithelialization. They were considered completely reepithelized when no exudate was noted, the participant reported no pain with exposure of the wound to ambient air and was completely devoid of Membracel coverage and hematic crusts.

CONTACTS AND LOCATIONS:
Overall Officials: Rosadelia M Carboni, Student, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No